CLINICAL TRIAL: NCT04891380
Title: Prehospital Use of a Ballistocardiographic Biosensor to Non-invasively and Invasive Pulse Contour Analysis to Monitor Hemodynamics and Blood Flow During Emergency Medicine Cases, a Prehospital Prospective Feasibility Study
Brief Title: BCG Biosensor and Non- and Invasive Monitoring During Emergency Medicine Cases, a Prospective Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian Telemedicine (Unknown); Kopera Norway (Unknown); Edwards Medical (Unknown); Stryker Medical (Industry); University of Bilbao (Unknown); University of Stavanger (Other)
Responsible Party: Principal Investigator, Lars Wik, Principal Investigator, Oslo University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 205218
Record Dates: First submitted 2021-05-04; First posted 2021-05-18 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Cardiac Arrest, Out-Of-Hospital; Hypotension and Shock
Keywords: blood flow; rosc; cpr process; invasive blood pressure; cardiac output
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Hypotension; Shock | interventions — Hypotension, Controlled

STUDY DESIGN:
Intervention Model Description: All patients who meet the inclusion criterias will be eligiable.
Masking Description: It is impossible to mask since the devices used must be put on and operated by the responsible crew.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cardiac arrest patients (Other): Cardiac arrest patients receiving cardiopulmonary resuscitation with LUCAS 2 Active Decompression 2.
  Interventions: Device: LUCAS 2 Active Decompression 2
- Hypotension (Other): Patients developed or may develope hypotension of non traumatic origin.
  Interventions: Other: Hypotension
- Intensive care patient transport (Other): Patients who are transported from one intensive department to another.
  Interventions: Other: Intensive care transport
- LUCAS 2 Active Decompression (Other): The hemodynamic measurements of the cardiac arrest patients in the present study will be compared with the hemodynamic measurements achieved in the previous study NCT02479152.
  Interventions: Device: LUCAS 2 Active Decompression 2

INTERVENTIONS:
Device: LUCAS 2 Active Decompression 2 — Chest compression with active decompression of the chest. Measurement of physiological parameters.
  Other Names: FloTrac ™; BCG; Cerebral oximetry
  Arms: Cardiac arrest patients; LUCAS 2 Active Decompression
Other: Hypotension — measurement of physiological parameters
  Arms: Hypotension
Other: Intensive care transport — Measurement of physiological parameters
  Arms: Intensive care patient transport

SUMMARY:
In a out of hospital emergency medicine study the investigators will measure hemodynamic effects of implemented treatments for patients with cardiac arrest, hypotension, and intensive care transports. The investigators will use both non-invasive and invasive measuring technology to measure this. Ballistocardiographic biosensors are introduced together with more advanced non-invasive and invasive measurements such as invasive arterial blood pressure with cardiac output calculation and saturation cerebral tissue oxygenation (SctO2). During treatment of cardiac arrest patients the investigators will use a new LUCAS 2 Active Decompression device (LUCAS 2 AD2) and measure different hemodynamic variables.

DETAILED DESCRIPTION:
Pre-hospital monitoring of vital signs has documented to increase survival. Especially advanced multi-monitoring units have shown to have this impact but they are demanding in use. Low blood pressure/blood flow are frequent in emergency medicine cases and diagnosed by combining clinical evaluation (breathing, circulation, neurology) with biosensor measures of vital signs. Examples of biosensors are ECG, Ballistocardiographic (BCG), End Tidal CO2 (EtCO2), pulse oximetry (SpO2), saturation cerebral tissue oximetry (SctO2), transthoracic impedance (TTI), and invasive arterial pressure measurements such as pulse contour analysis for cardiac output measures. The gold standard for blood flow measurement is cardiac output [Cardiac Output (CO), volume of blood pumped by the heart pr. minute as the product of stroke volume (SV) and heart rate]. Cardiac output may be measured by invasive (thermodilution, Fick method) or noninvasively techniques [oesophageal Doppler, transoesophageal echocardiography, lithium dilatation cardiac output, pulse contour cardiac output (PICCO, Pulse Cardiac Output system, FloTrac ™), partial CO2 rebreathing, thoracic electrical bioimpedance. Pulse contour analysis is based on that the area under the systolic part of the arterial pressure waveform is proportional to the stroke volume (SV). This may limit the optimal goal for monitoring adequately several emergency medicine cases. There is, therefore, a need to develop and evaluate biosensor devices in these situations. BCG biosensors have been introduced and have documented to be useful in monitoring noninvasively vital signs but they have not been used in acute emergency medicine. It has been documented a correlation (r2=0.85) between BCG biosensor and cardiac output measured by Doppler echocardiogram. The biosensor record very subtle rhythmic movements on the patient skin (abdomen and/or neck) and shows a graph which is presented based on filters and custom-made algorithms as continuous hemodynamic variables (heart- and respiration-rates, heart rate variability, and relative stroke volume). BCG piezoelectric biosensors (BGPS) are easy to put on the patient, non-invasive, light (grams), small (2 x 2 cm), and costs are low. They support live streaming with automatic downloads of data. For most other measuring devices this must be done manually post event. With limited time of education and training all personnel prehospitally can deploy the biosensor over the carotid or abdominal aorta. Based on pilots and a validation study comparing two BCG biosensors (accelerometer and piezoelectric) with measures performed by present clinical practise the piezoelectric biosensor is best for use in situations where measures must be instant. In the same validation study, the investigators documented that pulse contour analysis with the latest software upgrade of FloTrac™ system worked well compared with Doppler echocardiography (manuscript in progress, ClinTrialGov). Studies have validated the efficacy of FloTrac ™ with pulmonary artery catheter and found different results. A review article concluded that FloTrac ™ has the possibility to increase patient safety in relation to perioperative hemodynamic monitoring. A comparison of simultaneous Stroke Volume (SV) and Cardiac Output measurements by echocardiography and FloTrac ™ were done in ten mechanically ventilated intensive care patients and showed a correlation between them (SV, y = 0.9545x + 3.3, R2 = 0.98 and for CO, y = 0.9104x + 7.7074, R² = 0.97). Therefore, it is indicated to use this biosensor for out of hospital cases. Although pulse contour analysis is an invasive method, the investigators have experience with invasive arterial access in the doctor car that respond to emergency cases in Oslo since invasive monitoring is the standard.

In a pre-hospital observational study performed by the doctor manned car (119-unit) in Oslo and Akershus, the investigators will compare and document (correlations, sensitivities, specificities) biosensor measures to current gold standard measures during cardiopulmonary resuscitation (CPR), hypotension, and intensive care transports. This challenges the current practice because most pre-hospital units responding to emergency medicine cases do not have alternatives to advanced measures. Therefore, the patient is not monitored well enough in addition to that they seldom receive instant guidance according to the effect of treatment. The investigators approach is novel and innovative since it has never been done but the investigators study group have recent experience with performing similar advanced clinical monitoring studies prehospitally. There is a potential that more pre-hospital units will deliver better monitoring and care to more patients with these non- and invasive approaches. Ultimately, better healthcare will be provided.

The data captured for the cardiac arrest patients will be compared with data from NCT02479152.

If the current project is successful, the investigators plan to implement this technology in a larger scale and may then be able to study potentially improved survival and morbidity rates with sufficient statistical power in future studies.

ELIGIBILITY:
Inclusion Criteria:

* Non-traumatic cardiac arrest, hypotension, intensive care transport where an attempt of resuscitation and treatment is considered appropriate in patients age ≥18 years.

Exclusion Criteria:

* Age <18 years.

  * Traumatic cardiac arrest
  * Known pregnancy (can be included in the hypotension group)
  * Victim not to be resuscitated (DNR orders)
  * Internals in prison
  * Included once in the study already
  * Patients too small for LUCAS 2-AD2 < 18.5 cm chest height
  * Patient too big for LUCAS 2-AD2 > 27.3 cm chest height
  * Chest or upper abdomen surgery (Large scars on the chest, only in the CPR group.
  * Sustained Restoration Of Spontaneous Circulation (ROSC) occurring before the LUCAS 2-AD2 can be applied to the patient, such that further CPR is not needed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2024-01-03 (Actual); Study Completion 2024-01-03 (Actual)

PRIMARY OUTCOMES:
End tidal partial pressure of CO2 (EtCO2). | Day 1
  Physiologic parameter EtCO2 is measured in the endotracheal tube.

SECONDARY OUTCOMES:
Saturation of cerebral tissue oxymetry (SctO2) | Day 1
  Physiologic parameter SctO2 is measured non invasive with Near Infrared spectroscopy.
Ballistocardiographic measurement of stroke volume in the aorta | Day 1
  Physiologic parameter Ballistocardiography measure non invasive the pulse or chest compression wave generated through the aorta.
Blood pressures | Day 1
  Physiologic parameters of Invasive measurement of systolic, diastolic and mean arterial blood pressures.
Cardiac output | Day 1
  Physiologic parameter to measure blood flow generated by the heart with the use of pulse contour waveform technology.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Wik, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Please Select, Norway

IPD SHARING:
Plan to Share IPD: Yes
Sharing will be done using an approved data sharing program
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all patients included. Available for 36 months
Access Criteria: Data will be shared with University of Bilbao and Stavanger, Stryker, and Edwards